CLINICAL TRIAL: NCT00090467
Title: Biochemical and Genetic Markers of Hypertension in Women
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Howard D. Sesso, ScD, MPH, Associate Epidemiologist, Brigham and Women's Hospital
Other Study IDs: 1267; R01HL075455-01 (NIH)
Record Dates: First submitted 2004-08-26; First posted 2004-08-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Cardiovascular Diseases; Hypertension; Heart Diseases; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Heart Diseases; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
To investigate biochemical and genetic markers of inflammation and endothelial dysfunction as determinants of hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension affects up to 50 million Americans, and is a major risk factor for cardiovascular disease and other health outcomes. Among Black women, hypertension is more prevalent, less well controlled by treatment, and has more damaging health outcomes versus Whites for reasons still unclear. While several lifestyle and dietary factors are associated with hypertension, relevant biochemical and genetic markers remain less well studied

DESIGN NARRATIVE:

This is a nested case-control study of incident hypertension in 800 case-control pairs (400 each of white and black women, totaling 1,600 women). Data will be used from the Women's Health Initiative Observational Study (WHI-OS), a cohort of 93,676 ethnically diverse postmenopausal women aged 50 to 79 years with extensive clinical and questionnaire data. Three hypotheses will be tested. First, the investigators will assess whether markers of inflammation - C reactive protein (CRP), interleukin-6 (IL-6), IL-1-8, tumor necrosis factor (TNF) receptor 2, soluble intercellular adhesion molecule-1 (slCAM-1), and metalloproteinase-9 (MMP-9) - are associated with the risk of hypertension in White and Black women. Second, they will examine six novel polymorphisms linked to the above inflammatory biomarkers - the CRP, IL-6, IL-1-beta, TNF-a, slCAM-1, and MMP-9 genes- and two other polymorphisms related to inflammation and the metabolic syndrome- the adiponectin and PPAR-y2 genes - for their potentially important associations with the risk of hypertension. Third, they will comprehensively evaluate important single-nucleotide polymorphisms in the above genes and examine associations between common haplotypes and hypertension risk in White and Black women, using state-of-the art genotyping technology and statistical methods. Power is excellent; for each biochemical marker, they have 80% power to detect a trend across quintiles for a relative risk (RR) of hypertension, comparing the fifth versus first quintiles, of 1.49 for analyses of 800 case-control pairs and 1.74 for analyses of 400 case-control pairs. For each genetic marker, they have 80% power to detect an additive effect of an allele for a RR of hypertension of 1.36 for 800 case-control pairs and 1.57 for 400 case-control pairs.

ELIGIBILITY:
We included White and Black WHI-OS participants aged <70 years, and excluded women with any baseline history of hypertension (via self-report, measured BP, or medication use), non-melanoma cancer, myocardial infarction, revascularization procedures, congestive heart failure, angina pectoris, or stroke. Further, women developing myocardial infarction or stroke, or dying from coronary heart disease or stroke during follow-up were excluded. Only for potential hypertension cases, women with revascularization procedures, congestive heart failure, angina pectoris, or non-melanoma cancer prior to or <30 days after the diagnosis of hypertension were also excluded. Finally, we excluded women with inadequate bloods or who refused to participate in a genetic study.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women's Health Initiative Observational Study (WHI OS)
Sampling Method: Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2004-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incident hypertension | Median follow-up of 5.9 years

CONTACTS AND LOCATIONS:
Overall Officials: Howard D Sesso, ScD, MPH, Principal Investigator — Brigham & Women"s Hospital